CLINICAL TRIAL: NCT01161420
Title: Effects of the Inspire Implantable Nerve Stimulation System on Obstructive Sleep Apnea
Brief Title: Stimulation Therapy for Apnea Reduction (Www.theSTARtrial.Com)
Acronym: STAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Inspire Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Inspire 4
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: tongue; surgery; neurostimulation; hypoglossal nerve; upper airway stimulation
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inspire Therapy (Experimental): Inspire Upper Airway Stimulation System, is a permanent, implantable therapy device, which consists of three implantable components: IPG, stimulation lead, and a sensing lead. In additional the patient receives a remote to activate the therapy.
  Interventions: Device: Inspire Upper Airway Stimulation System

INTERVENTIONS:
Device: Inspire Upper Airway Stimulation System — Inspire Upper Airway Stimulation System, is a permanent, implantable therapy device, which consists of three implantable components: IPG, stimulation lead, and a sensing lead. In additional the patient receives a remote to activate the therapy.
  Other Names: Inspire; UAS; Inspire Therapy

SUMMARY:
The purpose of this clinical trial is to demonstrate long-term safety and efficacy of the Inspire system. The Inspire Upper Airway Stimulation (UAS) therapy is intended to treat moderate-to-severe obstructive sleep apnea by improving airway patency through stimulation of the hypoglossal nerve. Study objectives include demonstrating that the Inspire system improves key indices of sleep apnea in a pre-specified percentage of patients.

DETAILED DESCRIPTION:
The STAR trial is a multicenter, prospective trial that includes a randomized controlled therapy withdrawal study. The primary and secondary endpoint data were collected during an in-laboratory sleep study 12 months after the device implant and were compared against the baseline sleep studies. Following the 12-month visit, 46 consecutive responding subjects were randomized 1:1 to either a therapy maintenance group (ON group) or a therapy withdrawal group (OFF group). A subsequent sleep study of the two randomized groups was conducted and results were compared between the two groups. In addition, quality of life questionnaires were administered at baseline and at the 12-month visit to further assess the effectiveness of Inspire therapy.

The STAR trial was conducted at 15 clinical sites in the United States and 7 in Europe. Of the 126 implanted subjects in the STAR trial, 87 or 69% were implanted in the United States. The remaining 39 subjects or 31% were implanted in Europe.

The STAR trial subjects were evaluated prior to implant to ensure the following: 1) that their pre-implant AHI (as scored during an in-laboratory sleep study prior to implant) was between 20 and 50 events per hour, 2) that any AHI contribution from central or mixed sleep apnea was less than 25%, 3) that subjects did not have primarily lateral OSA (defined as limited sleep apnea when lying on their side), and 4) that the subjects did not have a complete concentric collapse at the level of the soft palate while observed during a drug-induced sleep endoscopy (DISE).

After successful pre-implant screening, the subjects were implanted with the Inspire system. The subjects were allowed to recover for 1 month following surgery, at which time a second in-laboratory sleep study was conducted without activating the Inspire device. The results of this 1-month sleep study were averaged with the results of the pre-implant sleep study, and the average is defined as the subject's baseline.

The Inspire device is programmable in order to optimize a subject's response to therapy. The initial device settings are programmed in an office setting. Additional adjustments are made during an overnight sleep study whereby real time review of the polysomnogram (PSG) is available to aid in device setting adjustments during the 2 and 6-month visit.

At the 12-month in-laboratory sleep study, no device adjustments were allowed as this sleep study was the primary endpoint sleep study. Furthermore, no device adjustments were allowed at the 13-month sleep study which was the randomized controlled therapy withdrawal sleep studies.

Blinding was not possible during the study since the stimulation therapy evokes a physiological response in the subjects. However, the primary endpoints were based on the objective measures of AHI and oxygen desaturation index (ODI) which were collected during an overnight sleep study using PSG. The sleep studies were all scored by an independent core lab in order to minimize assessment bias. Furthermore, the sleep study results, as well as all other clinical results, were 100% source data verified by the Inspire clinical monitoring team.

ELIGIBILITY:
Inclusion Criteria:

* Likely suffer moderate-to-severe OSA based on history and physical
* Have failed or have not tolerated CPAP treatment
* Willing and capable of providing informed consent
* Willing and capable to have stimulation hardware permanently implanted, and to use the patient programmer to activate the stimulation
* Willing and capable to return for all follow-up visits and sleep studies, including the evaluation procedures and filling out the questionnaires

Exclusion Criteria:

* Body Mass Index limits
* Surgical resection or radiation therapy for cancer or congenital malformations in the larynx, tongue, or throat
* Significant co-morbidities making the patient unable or inappropriate to participate in the trial

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 929 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quan Ni, Ph.D., Study Director — Inspire Medical Systems, Inc.
Locations (22):
- United States (15):
  - California Sleep Institute, Palo Alto, California
  - Clinical Research Group of St. Petersburg, Inc., St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - Advanced ENT, Atlanta, Georgia
  - Wayne State University / Detroit Medical Center, Detroit, Michigan
  - Borgess Research Institute, Portage, Michigan
  - North Memorial Medical Center, Maple Grove, Minnesota
  - St. Cloud ENT, Saint Cloud, Minnesota
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals / Case Western Reserve, Cleveland, Ohio
  - University of Pittsburgh Medical Center; Montefiore, Oakland, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sleep Medicine Associates of Texas, Dallas, Texas
  - Swedish Health Services, Seattle, Washington
  - Froedtert Memeorial Hospital, Milwaukee, Wisconsin
- Deparment of Pulmonology Head and Neck Surgery, Universitair Ziekenhuis Antwerpen, Antwerp, Belgium
- France (2):
  - Central Hospital University of Bordeaux, Bordeaux
  - Hospital Foch, Paris
- Germany (3):
  - Krankenhaus Bethanien Solingen, Solingen, DE
  - St. Franziskus Hospital, Cologne
  - Universitäts-HNO-Klinik Mannheim, Mannheim
- St. Lucas Andreas Ziekenhuis, Amsterdam, Netherlands

REFERENCES:
- [Derived] Johnson MD, Dweiri YM, Cornelius J, Strohl KP, Steffen A, Suurna M, Soose RJ, Coleman M, Rondoni J, Durand DM, Ni Q. Model-based analysis of implanted hypoglossal nerve stimulation for the treatment of obstructive sleep apnea. Sleep. 2021 Apr 27;44(44 Suppl 1):S11-S19. doi: 10.1093/sleep/zsaa269. PMID 33647987
- [Derived] Yu JL, Younes M. Relation between arousability and outcome of upper airway stimulation in the Stimulation for Apnea Reduction (STAR) Trial. J Clin Sleep Med. 2021 Apr 1;17(4):797-801. doi: 10.5664/jcsm.9050. PMID 33295277
- [Derived] Op de Beeck S, Wellman A, Dieltjens M, Strohl KP, Willemen M, Van de Heyning PH, Verbraecken JA, Vanderveken OM, Sands SA; STAR Trial Investigators. Endotypic Mechanisms of Successful Hypoglossal Nerve Stimulation for Obstructive Sleep Apnea. Am J Respir Crit Care Med. 2021 Mar 15;203(6):746-755. doi: 10.1164/rccm.202006-2176OC. PMID 32970962
- [Derived] Strollo PJ Jr, Soose RJ, Maurer JT, de Vries N, Cornelius J, Froymovich O, Hanson RD, Padhya TA, Steward DL, Gillespie MB, Woodson BT, Van de Heyning PH, Goetting MG, Vanderveken OM, Feldman N, Knaack L, Strohl KP; STAR Trial Group. Upper-airway stimulation for obstructive sleep apnea. N Engl J Med. 2014 Jan 9;370(2):139-49. doi: 10.1056/NEJMoa1308659. PMID 24401051
- See also: Click here for more information about the intervention — http://www.inspiresleep.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 10 Nov 2010 and 15 Feb 2012, 25 clinical sites enrolled 929 subjects into the study. A total of 803 subjects were withdrawn from the study as they were not eligible and did not receive an implant.126 subjects from 22 clinical sites were implanted the UAS system (3 clinical sites enrolled subjects but did not attempt or implant a device).
Pre-assignment Details: 126 subjects were implanted with the Inspire therapy. At 12 months, the first 46 therapy responders were randomized 1:1 to either therapy ON (maintenance) or therapy OFF (withdrawal) for one week. Those who were in the withdrawal group returned to full therapy after one week of therapy being turned off.
Groups:
- Inspire Therapy: 126 subjects were implanted with Inspire therapy
Period: Inspire Therapy
Arm/Group | Inspire Therapy
Started | 126
Completed | 124
Not Completed | 2
Period: Withdrawal Study - Maintenance
Arm/Group | Inspire Therapy
Started | 23
Completed | 23
Not Completed | 0
Period: Withdrawal Study - Withdrawal
Arm/Group | Inspire Therapy
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Sample size was estimated using SAS V9.2 software using the two-sided, two-sample t-test for normal population.
Groups:
- Inspire Therapy: Study subjects continue to use Inspire therapy
  Inspire Upper Airway Stimulator: The stimulator is surgically positioned subcutaneously near the clavicle in the upper chest, and connects to a stimulation lead (around a hypoglossal nerve) and a sensing lead (in the chest). The stimulation contracts a patient's upper airway muscles to maintain airway patency, with the intent to keep the airway open during inspiration.
Arm/Group | Inspire Therapy
Number analyzed (Participants) | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (10.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 110
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 105
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 122
  More than one race | 0
  Unknown or Not Reported | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 123
Region of Enrollment [Number; unit: participants]
  France | 2
  United States | 87
  Belgium | 4
  Netherlands | 22
  Germany | 11

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index
Description: Demonstrate at least a 50% responder rate at the 12-month follow-up visit. An Inspire therapy AHI responder was defined as a subject who experienced at least a 50% reduction in AHI from baseline and had an AHI of less than 20 at the 12-month follow-up.
Time Frame: 12 months
Measure: Number; unit: percentage of subjects responding
Groups:
- Inspire Therapy: Study subjects continue to use Inspire therapy; Inspire Upper Airway Stimulator: The stimulator is surgically positioned subcutaneously near the clavicle in the upper chest, and connects to a stimulation lead (around a hypoglossal nerve) and a sensing lead (in the chest). The stimulation contracts a patient's upper airway muscles to maintain airway patency, with the intent to keep the airway open during inspiration.
Arm/Group | Inspire Therapy
Number analyzed (Participants) | 126
percentage of subjects responding | 66 [9.3 to 23.6]

2. Primary Outcome: Oxygen Desaturation Index
Description: Demonstrate at least a 50% responder rate at the 12-month follow-up visit. An Inspire therapy ODI responder was defines as a subject who experienced at least a 25% reduction in ODI from baseline.
Time Frame: 12 months
Measure: Number; unit: percentage of subjects responding
Arm/Group | Inspire Therapy
Number analyzed (Participants) | 126
percentage of subjects responding | 75 [13.9 to 15.7]

3. Primary Outcome: Safety
Description: The primary safety objective of this pivotal trial was to evaluate safety via a description of all reported adverse events. Per the IDE-approved protocol, no formal statistical hypothesis was tested as part of the safety assessment.
Time Frame: 12 months
Measure: Number; unit: Events Reported
Groups:
- All Subjects: 126 implanted study subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 126
Events Reported | 494

4. Secondary Outcome: AHI for the Randomized Controlled Therapy (RCT) Withdrawal Study
Description: The AHI difference between the 12-month PSG study and the 13-Month PSG study in the therapy maintenance group will be compared to the AHI difference in the therapy withdrawal group. The objective was to demonstrate that AHI increase in the therapy withdrawal group (therapy=OFF) is greater than any AHI change in the active therapy group (therapy=ON). AHI is the number of apneas or hypopneas recorded during a sleep study per hour of sleep; this is calculated by dividing the number of AHI events by the number of hours of sleep.
Time Frame: 12 Months
Population: The first 46 responders to the Inspire therapy at 12 months were randomized 1:1 to either the Therapy Maintenance Group (ON) or the Therapy Withdrawal Group (OFF). A subsequent sleep study of the two randomized groups was conducted and results were compared between the two groups.
Measure: Mean (95% Confidence Interval); unit: events per hour
Groups:
- Maintenance: Twenty-three (23) patients were in the therapy maintenance (ON) group
- Withdrawal: Twenty-three (23) patients were in the therapy withdrawal (OFF) group.
Arm/Group | Maintenance | Withdrawal
Number analyzed (Participants) | 23 | 23
events per hour | 12.0 [9.3 to 23.6] | 16.4 [9.3 to 23.6]

5. Secondary Outcome: Modified Intent to Treat - AHI Responder Rate for All Implanted Subjects
Description: The intent-to-treat (ITT) analysis for the primary endpoint included all patients who underwent an implant. A modified ITT analysis was conducted to include the subjects who did not completed the 12-month follow-up sleep study also. The ITT analysis was to calculate the AHI responder rate based on the subjects included in the analysis as described below. An Inspire therapy AHI responder was defined as a subject who experienced at least a 50% reduction in AHI from baseline and had an AHI of less than 20 at their last visit.
  The following subjects were included:
  * All implanted subjects who had AHI data collected at both baseline and 12-months follow-up.
  * All implanted subjects who had baseline data but no 12-month data, and had their last data values carried forward, provide they had a least 6-month AHI data.
  * Any implanted subject who did not have 12-month data available due to therapy failure (e.g., study withdrawal will be included in the analsys as a treatment failure.
Time Frame: 12 months
Population: Implanted subjects
Measure: Number; unit: Number of subjects responding to therapy
Groups:
- Inspire Therapy: 126 subjects implanted with Inspire therapy
Arm/Group | Inspire Therapy
Number analyzed (Participants) | 126
Number of subjects responding to therapy | 83

6. Secondary Outcome: Change in FOSQ From Baseline to 12 Months
Description: The Functional Outcomes Sleep Questionnaire (FOSQ) is a validated instrument that assesses the effect of a subject's daytime sleepiness on activities of ordinary living. It is a quality of life measure that is commonly used in the clinical evaluation and management of OSA. This self-administered instrument consists of 30 questions divided into 5 domains: activity level, vigilance, intimacy, general productivity and social outcome. Scores range from 5 to 20, with higher scores indicating greater functioning. Change in FOSQ was calculated by subtracting the baseline score from the 12-month score.
Time Frame: Baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Inspire Therapy: 126 subjects completed the baseline questionnaire, however 123 study subjects completed the 12-month questionnaire; two subjects did not completed this questionnaire and one subject expired.
Arm/Group | Inspire Therapy
Number analyzed (Participants) | 123
units on a scale | 2.9 [2.4 to 3.5]

7. Secondary Outcome: Change Epworth Sleepiness Scale (ESS) From Baseline to 12 Months
Description: The Epworth Sleepiness Scale (ESS) is a validated instrument that rates a subject's daytime sleepiness. Like the FOSQ, it is a quality of life measure that is commonly used in clinical evaluation and management of OSA. Scores range from 0 to 24, with lower scores indicating greater functioning. An ESS score of less than 10 is considered to be the cutpoint for normal subjective sleepiness.
Time Frame: Baseline and 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Inspire Therapy
Number analyzed (Participants) | 123
units on a scale | 4.7 [3.8 to 5.5]

8. Secondary Outcome: Percentage Sleep Time at SaO2 < 90%
Description: The percentage of time spent with oxygen saturation below 90% has been an increasingly utilized surrogate for morbidity risk in sleep apnea populations.
  The SaO2 secondary endpoint in this study was determined by the time below an SaO2 level of 90% during the 12-month PSG study compared to that at baseline (average of screening and 1-month PSG studies). The objective was to demonstrate a decrease in the percentage of sleep time with an SaO2 level below 90% at 12 months.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: Percentage of Sleep Time SaO2 <90%
Groups:
- Inspire Therapy: 126 subjects were implanted with Inspire therapy; 124 subjects completed this visit (two expired prior to the 12-month visit).
Arm/Group | Inspire Therapy
Number analyzed (Participants) | 124
Percentage of Sleep Time SaO2 <90% | 2.5 (11.1) [0.6 to 4.5]

ADVERSE EVENTS:
Time Frame: For the submission adverse events were collected from 10 November 2010 to data cut-off of 12 February 2012. Adverse events continue to be collected for long-term follow-up.
Groups:
- Inspire Therapy: This pivotal trial was to evaluate safety via a description of all reported adverse events. Per the IDE-approved protocol, no formal statistical hypothesis was tested as part of the safety assessment.
Arm/Group | Inspire Therapy
Serious Adverse Events (participants affected / at risk) | 13/126
Other Adverse Events (participants affected / at risk) | 107/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inspire Therapy (N=126)
Device Revision - resuture to secure IPG (Surgical and medical procedures) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2) — pre-existing or independent condition unrelated to Inspire procedure or therapy.
Death (Cardiac disorders) | 1 (1) — pre-existing or independent condition unrelated to Inspire procedure or therapy.
Chest Pressure and/or Pain (Cardiac disorders) | 2 (2) — pre-existing or independent condition unrelated to Inspire procedure or therapy.
Recurring Syncope (Surgical and medical procedures) | 1 (1) — pre-existing or independent condition unrelated to Inspire procedure or therapy.
Coronary Artery Disease (Cardiac disorders) | 1 (1) — pre-existing or independent condition unrelated to Inspire procedure or therapy.
Rotator Cuff Injury (Injury, poisoning and procedural complications) | 1 (1) — pre-existing or independent condition unrelated to Inspire procedure or therapy.
Knee Injury (Injury, poisoning and procedural complications) | 1 (2) — pre-existing or independent condition unrelated to Inspire procedure or therapy.
Acute Entercolitis (Gastrointestinal disorders) | 1 (1) — pre-existing or independent condition unrelated to Inspire procedure or therapy.
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 1 (1) — pre-existing or independent condition unrelated to Inspire procedure or therapy.
Heart Catheter Procedure (Cardiac disorders) | 1 (1) — pre-existing or independent condition unrelated to Inspire procedure or therapy.
Accident (Injury, poisoning and procedural complications) | 1 (1) — pre-existing or independent condition unrelated to Inspire procedure or therapy.
Hernia (Injury, poisoning and procedural complications) | 1 (1) — pre-existing or independent condition unrelated to Inspire procedure or therapy.
Entercolitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inspire Therapy (N=126)
Events specifically related to an incision (Surgical and medical procedures) | 32 (45) — Since the Inspire device is implanted under general anesthesia and requires three skin incisions, several types of AEs can be expected with this type of surgical procedure.
Post-operative discomfort independent of any surgical incision (Surgical and medical procedures) | 31 (39) — The events reported in this category are common post-operative experiences from surgery such as pain, numbness, swelling or other post-operative discomfort that was not related to a specific surgical incision.
Temporary tongue weakness (Surgical and medical procedures) | 23 (35) — The events reported in this category describe a temporary tongue weakness as evidenced by tongue numbness, tongue weakness or reduction in movement, tongue pain or discomfort, minor effect on speech, or swelling in the area.
Intubation Effects (Surgical and medical procedures) | 15 (18) — All subjects were intubated during the surgical procedure, and therefore it was expected that subjects may experience the common effects of intubation, including sore throat, swallowing discomfort, or general soreness.
Post-op Headache (Nervous system disorders) | 8 (8) — There were 8 reports of a post-implant headache in 8 (6%) subjects. All 8 events have been fully resolved with medication (5), medication and massage/acupuncture (1), or no intervention (2).
Other post-op symptoms (Surgical and medical procedures) | 14 (22) — Fourteen (11%) subjects experienced a total of 22 events of post-operative symptoms including nausea, vomiting, drug reactions or miscellaneous pain or body soreness.
Procedure related Infection (mild or moderate) (Infections and infestations) | 1 (1) — Procedure-related infections are categorized as mild or moderate (within 0-30 days post-procedure).
Discomfort due to electrical stimulation (General disorders) | 42 (66) — The reports of discomfort due to the upper airway stimulation includes tongue pain, tongue movement limitations, neck/jaw discomfort or patient waking up due to stimulation strength.
Tongue abrasion (General disorders) | 20 (23) — During the STAR trial, subjects reported symptoms of a sore tongue or tongue discomfort, including several with visible abrasions.
Mouth dryness (General disorders) | 9 (9) — Mouth dryness is often associated with OSA due to subject having their mouth open during the night.
Mechanical pain associated with presence of device (General disorders) | 6 (6) — Six (5%) subjects experienced 6 events resulting from discomfort or pain associated with the presence of the device, most commonly associated with the IPG.
Temporary internal device usability or functionality complaint (Investigations) | 8 (9) — There were 9 adverse events reported where the cause was attributed to the operation of the Inspire system in 8 (6%) subjects.
Temporary external device usability or functionality (Investigations) | 3 (3) — There were 3 events related to the operation of the external components and in all 3 cases, this was attributed to the subject's use of the patient programmer.
Other acute symptoms (Surgical and medical procedures) | 14 (18) — This device-related adverse event code was created to include various event descriptions such as headaches, coughing, choking, dysphagia and speech.
Device related infection (Infections and infestations) | 1 (1)
Abdominal incisional pain (General disorders) | 1 (1)
Abdominal pain/faecal incontinence (Gastrointestinal disorders) | 1 (1)
Abnormal pap smear/HPV (Reproductive system and breast disorders) | 1 (1)
Abnormal x-ray (General disorders) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 1 (1)
Acute gastro-enteritis (Gastrointestinal disorders) | 1 (1)
Acute prostatitis (Reproductive system and breast disorders) | 1 (1)
Allgeric reaction to Diamox (Immune system disorders) | 1 (1) — Allergic reaction to Diamox
Allergic reaction to post-op antibiotics (Immune system disorders) | 1 (1)
Anxiety (Nervous system disorders) | 3 (3)
Awakening from sleep gasping for air (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient calling and describes awakening from sleep with a sense of gasping for air. She reports experiencing this in the past when she was not adaquately using her CPAP prior to implant
Back ache (Musculoskeletal and connective tissue disorders) | 1 (1) — lateral
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Benign fibrous papule and chronic folliculitis (Infections and infestations) | 1 (1)
Bilateral swelling of neck (General disorders) | 1 (1)
Blood in ejaculate (Reproductive system and breast disorders) | 1 (1)
Blood in sputum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bone spurs (Musculoskeletal and connective tissue disorders) | 1 (1)
BPH (Reproductive system and breast disorders) | 1 (1)
Broken teeth (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Burning, pinching, mildly tender at IPG site (General disorders) | 1 (1) — Baseball moves
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient complaint of pain in chest after waking up. This occurs only if patient takes a deep breath. This complaint was also there before the implant and has had it for years. However patient had not notified this before the implant date.
Common cold (Respiratory, thoracic and mediastinal disorders) | 8 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cytomegalovirus (Immune system disorders) | 1 (1)
Depression (Immune system disorders) | 2 (2)
Device stimulation not felt during the night (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Difficulty voiding (Renal and urinary disorders) | 1 (1)
Dilated cardiomyopathy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Drowsiness after Zolpidem administration (General disorders) | 1 (1)
Drug reaction (Immune system disorders) | 1 (1)
Dry throat (General disorders) | 1 (1)
Dysphagia (General disorders) | 1 (1) — Likely postoperative edema, mild. History of a Schatzki Ring dilation in the past.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ear pain (General disorders) | 1 (1) — Ear infection
Elevated triglycerides & blood sugar (Blood and lymphatic system disorders) | 1 (1) — Hyperglycemia - unspecified Hypertriglycerides - unspecified
Enlarged lymphnodes (Immune system disorders) | 1 (1) — possible viral infection
Fatigue related to B12 deficiency (General disorders) | 1 (1)
Patient fall (General disorders) | 4 (5) — Bicycle, ladder, general
Flu (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Grastic pain (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal discomfort with nausea and mild diarrhea (Gastrointestinal disorders) | 1 (1)
General malaise (General disorders) | 1 (1)
Generalized itching (General disorders) | 1 (1)
Generalized neuropathy (Nervous system disorders) | 1 (1)
GERD (Gastrointestinal disorders) | 1 (1)
GI Upset (Gastrointestinal disorders) | 1 (1)
Hangover symptoms with associated nausea and vomiting (General disorders) | 1 (1)
Head cold (General disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 (1)
Herpes Zoster (Shingles) (Nervous system disorders) | 2 (2)
Hyperhidrosis (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Itchy right ear (General disorders) | 1 (1) — Otitis externa
Impacted wisdom tooth (Musculoskeletal and connective tissue disorders) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1)
Infection of the throat (Infections and infestations) | 1 (1) — Intercurrent Infection (Viral)
Inflammation (General disorders) | 1 (1) — Light inflammation of the wound in the neck. Probably caused by shaving.
Insomnia (General disorders) | 3 (3)
Jolting sensation of whole body (General disorders) | 1 (1) — brief jerk/jolt of whole body and sense of falling immediately upon drifting to sleep with naps during the day. Not at night with use of Inspire therapy
Knee pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Left hip/groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left middle finger smashed (General disorders) | 1 (1)
Low grade headache (General disorders) | 1 (1)
Lower back muscle pull (Musculoskeletal and connective tissue disorders) | 1 (1)
Mould infection (mouth) (General disorders) | 1 (1) — Candida infection in mouth.
Nasal allergies (Immune system disorders) | 1 (1)
Nasal congestion (General disorders) | 1 (1)
Nightmares (General disorders) | 1 (1)
Non-cardiac chest pain (Nervous system disorders) | 1 (1) — anxiety
Obesitas (General disorders) | 1 (1)
Otitis media with effusion (Ear and labyrinth disorders) | 1 (1) — Patient reports L ear fullness with worsening allergies.
Pain after tooth extraction (General disorders) | 1 (1)
Pain below right shoulder (General disorders) | 1 (1)
Pain in esophagus (General disorders) | 1 (1)
Pain in right ear (General disorders) | 1 (1) — Slight infection
Pain in shoulder (General disorders) | 1 (1)
Painful back muscles (General disorders) | 1 (1)
Painful big toe (General disorders) | 1 (1) — bruised big toe
Painful hip (Musculoskeletal and connective tissue disorders) | 1 (1) — muscle strain
Painful right arm (Musculoskeletal and connective tissue disorders) | 1 (1) — muscle strain
Painful right index finger (Musculoskeletal and connective tissue disorders) | 1 (1) — flexor tendinitis
Personal and work related problems (General disorders) | 1 (1)
Pharyngitis (General disorders) | 2 (3)
Problems with jaw joint (General disorders) | 1 (1)
Rash (Immune system disorders) | 2 (2) — allergic reaction to penicillin
Prostatism (Reproductive system and breast disorders) | 1 (1)
Restless legs (Nervous system disorders) | 1 (1)
Right shoulder arm pain (General disorders) | 3 (3)
Right thigh hematoma (General disorders) | 1 (1)
Sciatic nerve aggravated (General disorders) | 1 (1)
Sinus infection (General disorders) | 3 (3)
Sinus/allergy symptoms (General disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Soft tissue pain; back/ribs (Musculoskeletal and connective tissue disorders) | 1 (1)
Stiff neck pain (General disorders) | 1 (1)
Stress (General disorders) | 2 (2)
Stuffy nose (General disorders) | 2 (2)
Submandibular gland pain (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
TBI with no LOC (General disorders) | 1 (1)
Throat ache (General disorders) | 1 (1)
Throat infection (General disorders) | 1 (1)
Throat pain (General disorders) | 1 (1)
Throat tightness (General disorders) | 1 (1)
Tinnitus (General disorders) | 2 (2)
Tongue biting (General disorders) | 1 (1)
Tongue hematoma (General disorders) | 1 (1)
Tongue pain (General disorders) | 1 (1)
Tooth ache (General disorders) | 1 (1)
Tooth infection (General disorders) | 1 (1)
Tooth removed (General disorders) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1)
Trigger fingers (General disorders) | 1 (1)
Type ll Diabetes (Endocrine disorders) | 1 (1)
Umbilical hernia (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Vaginal dermititis (Reproductive system and breast disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1)
Worsening arrhythmia - bigeminy (Cardiac disorders) | 1 (1)
Worsening occasional difficulty with speech (General disorders) | 1 (1) — Patient describes being "tongue tied" occasionally. States he has had this since TMJ surgery in 1994, but has noticed an increase in the last six months.
Worsening dry mouth (General disorders) | 1 (1)
Worsening urinary incontinence (Renal and urinary disorders) | 1 (1)
Worsening RLS (Nervous system disorders) | 1 (1)
Worsening sinusitis (Infections and infestations) | 1 (1)
Wound on top of thumb (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No